Prospective Monitoring of Angiotensin Receptor Blocker Neprilysin Inhibitor in Older Adults with Heart Failure and Frailty

February 11, 2021

NCT04743063

### STUDY PROTOCOL

Prospective Monitoring of Angiotensin Receptor Blocker Neprilysin Inhibitor in Older Adults with Heart Failure and Frailty

**Preparation or Update Date:** 

01/14/2021

# **Protocol Revision Summary**

| Date | Summary of Changes |
|------------|---------------------------------------------|
| 01/14/2021 | Protocol preparation for study registration |

### **BACKGROUND**

- 1. Angiotensin receptor blocker neprilysin inhibitor (ARNI) sacubitril/valsartan (Entresto (1))
  - a. Approved in July 7, 2015
  - b. Indication: HF with reduced ejection fraction
- 2. PARADIGM-HF trial; ARNI vs enalapril (2)
  - a. N=8442, follow-up 2.3 years
  - b. Composite of cardiovascular death and HF hospitalization: 21.8% vs 26.5%
  - c. Safety endpoints: hypotension (14.0% vs 9.2%), renal failure (3.3% vs 4.5%), hyperkalemia (16.1% vs 17.3%), angioedema (0.4% vs 0.2%)
- 3. 2017 ACC/AHA/HFSA guidelines for management of heart failure (3)
  - a. The clinical strategy of inhibition of the renin-angiotensin system with <u>ACE</u> inhibitors (Level of Evidence: A), OR ARBs (Level of Evidence: A), OR ARNI (Level of Evidence: B-R) in conjunction with evidence-based beta blockers, and aldosterone antagonists in selected patients, is recommended for patients with chronic HFrEF to reduce morbidity and mortality.
  - b. The use of ACE inhibitors is beneficial for patients with prior or current symptoms of chronic HFrEF to reduce morbidity and mortality (Level of Evidence: A). Although the use of an ARNI in lieu of an ACE inhibitor for HFrEF has been found to be superior, for those patients for whom ARNI is not appropriate, continued use of an ACE inhibitor for all classes of HFrEF remains strongly advised.
  - c. The use of ARBs to reduce morbidity and mortality is recommended in patients with prior or current symptoms of chronic HFrEF who are intolerant to ACE inhibitors because of cough or angioedema (Level of Evidence: A). <u>Head-to-head comparisons of an ARB versus ARNI for HF do not exist.</u> For those patients for whom an ACE inhibitor or ARNI is inappropriate, use of an ARB remains advised.
  - d. In patients with chronic symptomatic HFrEF NYHA class II or III who tolerate an ACE inhibitor or ARB, <u>replacement by an ARNI is recommended to further reduce morbidity and mortality</u> (Level of Evidence: B).

- e. ARNI should not be administered concomitantly with ACE inhibitors or within 36 hours of the last dose of an ACE inhibitor (Level of Evidence: B). Oral neprilysin inhibitors, used in combination with ACE inhibitors can lead to angioedema and concomitant use is contraindicated and should be avoided.
- f. ARNI should not be administered to patients with a history of angioedema (Level of Evidence: C).
- 4. 2021 ACC/AHA/HFSA focused update (4)
  - a. For patients with newly diagnosed Stage C HFrEF, a beta-blocker and an ACEI/ARB/ARNI should be started in any order. Each agent should be up-titrated to maximally tolerated or target dose. Initiation of a beta-blocker is better tolerated when patients are dry and an ACEI/ARB/ARNI when patients are wet.

### STUDY OVERVIEW AND DESIGN

- 1. Study aims: To emulate a prospective surveillance of the effectiveness and safety of ARNI vs a comparator (ARB) in older adults with HFrEF and different frailty status.
- 2. Data source(s): Data from 2014 up to 2020 will be used.
  - a. Medicare Database
  - b. Optum Database
  - c. MarketScan Research Database
- 3. Sequential cohort monitoring design (see Figure 1): The monitoring analysis will include 1) retrospective analysis of available data (2015-2017) at the time of first analysis (January 2021) and 2) prospective analysis of new data (2018-2020) as they become available to the researchers. Within each database, we will emulate biannual updating of data by creating a propensity score (PS)-matched cohort of new users every 6-month interval, beginning on the first marketing of ARNI (July 7, 2015-December 31, 2015, and 6-month intervals afterwards). Each sequential cohort will be followed for development of the outcomes of

interest. Outcome analysis will be performed at a pre-specified 6-month interval (prospective analysis). The surveillance will be performed by frailty status (frail vs non-frail) at the time of drug initiation. The results from each database will be pooled using fixed-effects meta-analysis (assuming low heterogeneity across the databases).

Figure 1. Schematic of sequential monitoring design



### STUDY POPULATION

- 1. Study population (see Figure 2) is created for each calendar interval.
- 2. Initiation of ARNI or comparator (ARB)
  - a. ARB: any of azilsartan, candesartan, eprosartan, Irbesartan, losartan, Olmesartan, telmisartan, valsartan
  - b. Index date (day 0): prescription fill from July 7, 2015

- 3. Assessment of eligibility (eligibility assessment window: [-365, 0] days) See Appendix for list of codes.
  - a. Continuous enrollment for medical and drug insurance (Part A, B, and D)
  - b. Diagnosis of HF (outpatient diagnosis x2 or inpatient x1)
  - c. Reduced EF (<45%) algorithm (5)
  - d. No prior use of ARNI or comparator (exposure wash-out window: [-365, -1] days)
  - e. No recent HF hospitalization, defined as HF diagnosis (Appendix) in the primary position in the inpatient dataset (outcome wash-out window: [-60, 0] days)
  - f. No recent nursing facility stay, defined as any of the following claims in [-60, 0] days
    - i. Place of service: 31 (skilled nursing facility), 32 (nursing facility), 33 (custodial care facility)
    - CPT codes: 99301, 99302, 99303, 99311, 99312, 99313, 99315, 99316,
       99379, 99380, G0066
  - g. Excluded if age <65 years or exposure to both drugs on day 0
  - h. Contraindication to either drug (exclusion assessment window: [-60, 0] days, unless specified otherwise)
    - i. Hypotension
    - ii. Chronic kidney disease stage IV or V or dialysis
    - iii. Acute kidney injury
    - iv. Hyperkalemia
    - v. Angioedema: [-beginning of data, 0] days
  - i. If a patient meets the above-mentioned eligibility criteria more than once, only the first record will be included.

Figure 2. Study design outline for comparative effectiveness and safety analysis



### **MEASUREMENTS**

- 1. Exposure to ARNI or comparator
  - a. ARNI: sacubitril/valsartan (Entresto)
  - b. ARB (comparator): any of azilsartan, candesartan, eprosartan, Irbesartan, losartan, Olmesartan, telmisartan, valsartan
  - c. Note: prior ACEI use (commonly used for hypertension and HFrEF) is allowed. This choice will resemble a clinic situation that involves switching from ACEI to ARB or to ARNI.
  - d. Exposure risk window and gap between treatments allowed: 7 days (primary analysis) or 14 days (sensitivity analysis)

#### 2. Outcomes

- a. Effectiveness endpoint:
  - i. Primary: a composite of all-cause death or HF hospitalization
    - Note cardiovascular death was not used because National Death Index data were only available up to 2016. Instead, all-cause death was used.
    - HF hospitalization is defined as HF diagnosis primary position in the inpatient dataset
  - ii. Secondary: individual components separately
- b. Safety endpoint:
  - i. Primary: a composite of SAE, defined as any hospitalization or ED visit due to diagnosis codes in the primary position:
    - hypotension
    - acute kidney injury/acute kidney failure
    - hyperkalemia
    - angioedema
  - ii. Secondary: individual components

#### 3. Covariates

- a. Sociodemographic information: age, sex, race, dual eligibility
- b. Diseases: Chronic Conditions Data Warehouse (CCW) chronic conditions (see Table 2), provided in the Medicare Beneficiary Summary File (first date of satisfying the claims-based algorithm for individual conditions is available; considered present if this date is earlier than the index date)
- c. Prescription drugs: ATC3 classes with prevalence threshold >1% in a representative
   Medicare sample
- d. Gagne combined comorbidity score (6)
- e. Claims-based frailty index (7): Frailty status will be defined as non-frail if <0.20 or frail if ≥0.20

**Table 2. CCW Chronic Conditions (8)** 

| Acquired Hypothyroidism | Chronic Kidney Disease |
|---|---|
| Acute Myocardial Infarction | Chronic Obstructive Pulmonary Disease |
| Alzheimer's Disease, Related Disorders, or<br>Senile Dementia | Depression |
| Anemia | Diabetes |
| Asthma | Glaucoma |
| Atrial Fibrillation | Hip / Pelvic Fracture |
| Benign Prostatic Hyperplasia | Hyperlipidemia |
| Cancer (any of the following): | Hypertension |
| Cancer, Colorectal | Ischemic Heart Disease |
| Cancer, Endometrial Cancer, Breast | Osteoporosis |
| Cancer, Lung | Rheumatoid Arthritis / Osteoarthritis |
| Cancer, Prostate | Stroke / Transient Ischemic Attack |
| Cataract | |

### STATISTICAL ANALYSIS

### Estimation of treatment effectiveness and safety within each database

- 1. PS-matched cohorts: Within each surveillance cohort by frailty status (frail vs non-frail), we will use logistic regression that estimates the probability of receiving the drug of interest as a function of sociodemographic characteristics, diseases, prescription drugs, comorbidity index, and frailty index. Note that PS model will be fit separately by frailty status. We will perform a 1:1 ratio nearest-neighbor PS matching, with a caliper of 0.2 of the standard deviation of the logit PS (9). We will evaluate balance in covariates using standard mean difference (<0.1 is considered adequate balance) within each surveillance cohort.
- 2. Primary analysis for effectiveness and safety: For time-to-event analysis of the effectiveness and safety endpoints, we will use Cox proportional hazards regression to estimate the hazard ratios (HR) and 95% confidence intervals (CI) by frailty status (frail vs non-frail). The follow-up will begin on day 1 and end on the day of development of the effectiveness or safety endpoints or the earliest of the following censoring events: switching or discontinuation of the study drug, death not due to the outcome of interest, disenrollment, and end of data period (see Figure 2). Proportional hazards assumptions will be checked using Schoenfeld residuals.
- 3. Subgroup analyses for primary effectiveness and safety endpoints will be conducted <u>by</u> <u>frailty status (frail vs non-frail)</u>:
  - a. age (65-74 years vs  $\geq$ 75 years)
  - b. sex
  - c. race (black or non-black)
  - d. dual eligibility for Medicaid
  - e. major multimorbidity burden/pattern (informed by latent class analysis)
  - f. dementia (CCW definition)
  - g. HF hospitalization status ( $\geq 2$  or  $\leq 2$  in the past year)

- 4. Secondary analyses will be conducted by frailty status (frail vs non-frail):
  - a. secondary endpoints (individual components of primary effectiveness and safety composite endpoints)
- 5. Sensitivity analysis for primary effectiveness and safety endpoints will be conducted <u>by</u> frailty status (frail vs non-frail):
  - a. "intention-to-treat" analysis with a maximum follow-up time of 1 and 2 years from the index date
  - b. exposure risk window or grace period of 14 days
- 6. Adjustment for multiple testing in detecting signal: We will use the maximum sequential probability ratio testing (maxSPRT) procedure to keep the overall type-1 error rate of 0.05. (10)

### Estimation of the pooled treatment effectiveness and safety

- 7. The treatment effect estimates from 3 databases will be combined using meta-analysis techniques. We will examine the heterogeneity of treatment effect using Cochrane Q statistics and I-square statistics. If there is no statistically significant evidence of treatment effect heterogeneity, we will use inverse probability fixed-effects model to pool the database-specific estimates. If there is significant treatment effect heterogeneity, we will use random-effects model.
- 8. Reporting of prospective monitoring results: When a statistically significant signal is detected from the pooled analysis for the primary endpoints of effectiveness or safety from pre-specified interim analysis or at the end of the data period (12/31/2020), the findings will be reported

### **REFERENCES**

- https://www.accessdata.fda.gov/drugsatfda\_docs/label/2019/207620s013lbl.pdf. U.S.
   Food and Drug Administration; 2021.
- 2. McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, et al. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014;371(11):993-1004.
- 3. Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE, Jr., Colvin MM, et al. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. Circulation. 2017;136(6):e137-e61.
- 4. Maddox TM, Januzzi JL, Allen LA, Breathett K, Butler J, Davis LL, et al. 2021 Update to the 2017 ACC Expert Consensus Decision Pathway for Optimization of Heart Failure Treatment: Answers to 10 Pivotal Issues About Heart Failure With Reduced Ejection Fraction. Journal of the American College of Cardiology.0(0).
- 5. Desai RJ, Lin KJ, Patorno E, Barberio J, Lee M, Levin R, et al. Development and Preliminary Validation of a Medicare Claims-Based Model to Predict Left Ventricular Ejection Fraction Class in Patients With Heart Failure. Circ Cardiovasc Qual Outcomes. 2018;11(12):e004700.
- 6. Combined Comorbidity Score for Claims Data [Internet]. Available from: https://www.drugepi.org/dope/software
- 7. Claims-Based Frailty Index [Internet]. 2020 [cited December 1, 2020]. Available from: <a href="https://dataverse.harvard.edu/dataverse/cfi/">https://dataverse.harvard.edu/dataverse/cfi/</a>.
- 8. Chronic Conditions Data Warehouse [Internet]. 2020. Available from: https://www2.ccwdata.org/web/guest/condition-categories/
- 9. Austin PC. Optimal caliper widths for propensity-score matching when estimating differences in means and differences in proportions in observational studies. Pharm Stat. 2011;10(2):150-61.

10. Brown JS, Kulldorff M, Chan KA, Davis RL, Graham D, Pettus PT, et al. Early detection of adverse drug events within population-based health networks: application of sequential testing methods. Pharmacoepidemiology and Drug Safety. 2007;16(12):1275-84.

| Acute kie | dnav ini | ing Dy | |
|---|---|---|---|
| | | ICD10 Description | ICD9 Description |
| I120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, unspecified, with chronic kidney disease stage V |
| 1120 | .0371 | kidney disease or end stage renal disease | or end stage renal disease |
| N170 | 5845 | Acute kidney failure with tubular necrosis | Acute kidney failure with lesion of tubular necrosis |
| N171 | 5846 | Acute kidney failure with acute cortical necrosis | Acute kidney failure with lesion of renal cortical necrosis |
| N172 | 5847 | Acute kidney failure with medullary necrosis | Acute kidney failure with lesion of renal medullary [papillary] necrosis |
| N178 | 5848 | Other acute kidney failure | Acute kidney failure with other specified pathological lesion in kidney |
| N179 | 5849 | Acute kidney failure, unspecified | Acute kidney failure, unspecified |
| N19 | 586 | Unspecified kidney failure | Renal failure, unspecified |
| Z4931 | V560 | Encounter for adequacy testing for hemodialysis | Encounter for extracorporeal dialysis |
| Angioed | | | |
| | | ICD10 Description | ICD9 Description |
| T783XX | | Angioneurotic edema, initial encounter | Angioneurotic edema, not elsewhere classified |
| T783XXI | V5889 | Angioneurotic edema, subsequent encounter | Other specified aftercare |
| T783XX | | Angioneurotic edema, sequela | Late effect of other and unspecified external causes |
| | | disease stage IV or V or dialysis Dx | Tropo p |
| | | ICD10 Description | ICD9 Description |
| E1021 | | Type 1 diabetes mellitus with diabetic nephropathy | Diabetes with renal manifestations, type I [juvenile type], uncontrolled |
| E1022 | 25041 | Type 1 diabetes mellitus with diabetic chronic kidney disease | Diabetes with renal manifestations, type I [juvenile type], not stated as uncontrolled |
| E1029 | 25041 | Type 1 diabetes mellitus with other diabetic kidney complication | Diabetes with renal manifestations, type I [juvenile type], not stated as uncontrolled |
| E1065 | | Type 1 diabetes mellitus with hyperglycemia | Diabetes with renal manifestations, type I [juvenile type], uncontrolled |
| E1121 | | Type 2 diabetes mellitus with diabetic nephropathy | Diabetes with renal manifestations, type II or unspecified type, uncontrolled |
| E1122 | | Type 2 diabetes mellitus with diabetic chronic kidney disease | Diabetes with renal manifestations, type II or unspecified type, not stated as uncontrolled |
| E1129 | | Type 2 diabetes mellitus with other diabetic kidney complication | Diabetes with renal manifestations, type II or unspecified type, not stated as uncontrolled |
| E1165 | 25042 | Type 2 diabetes mellitus with hyperglycemia | Diabetes with renal manifestations, type II or unspecified type, uncontrolled |
| E1321 | 25040 | Other specified diabetes mellitus with diabetic nephropathy | Diabetes with renal manifestations, type II or unspecified type, not stated as uncontrolled |
| E1322 | 25040 | Other specified diabetes mellitus with diabetic chronic kidney disease | Diabetes with renal manifestations, type II or unspecified type, not stated as uncontrolled |
| E1329 | 25040 | Other specified diabetes mellitus with other diabetic kidney complication | Diabetes with renal manifestations, type II or unspecified type, not stated as uncontrolled |
| I120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic kidney disease or end stage renal disease | Hypertensive chronic kidney disease, unspecified, with chronic kidney disease stage V or end stage renal disease |
| I129 | 40390 | Hypertensive chronic kidney disease with stage 1 through<br>stage 4 chronic kidney disease, or unspecified chronic kidney<br>disease | Hypertensive chronic kidney disease, unspecified, with chronic kidney disease stage I through stage IV, or unspecified |
| I130 | | Hypertensive heart and chronic kidney disease with heart failure and stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| I1310 | 40490 | Hypertensive heart and chronic kidney disease without heart failure, with stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive heart and chronic kidney disease, unspecified, without heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| I1311 | 40492 | Hypertensive heart and chronic kidney disease without heart failure, with stage 5 chronic kidney disease, or end stage renal disease | Hypertensive heart and chronic kidney disease, unspecified, without heart failure and with chronic kidney disease stage V or end stage renal disease |
| I132 | 40493 | Hypertensive heart and chronic kidney disease with heart failure and with stage 5 chronic kidney disease, or end stage renal disease | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and chronic kidney disease stage V or end stage renal disease |
| N181 | 5851 | Chronic kidney disease, stage 1 | Chronic kidney disease, Stage I |
| N182 | 5852 | Chronic kidney disease, stage 2 (mild) | Chronic kidney disease, Stage II (mild) |
| N183 | 5853 | Chronic kidney disease, stage 3 (moderate) | Chronic kidney disease, Stage III (moderate) |
| N184 | 5854 | Chronic kidney disease, stage 4 (severe) | Chronic kidney disease, Stage IV (severe) |
| N189 | 5859 | Chronic kidney disease, unspecified | Chronic kidney disease, unspecified |
| N250 | 5880 | Renal osteodystrophy | Renal osteodystrophy |
| N251 | 5881 | Nephrogenic diabetes insipidus | Nephrogenic diabetes insipidus |
| N2581<br>N2589 | 58881<br>58889 | Secondary hyperparathyroidism of renal origin Other disorders resulting from impaired renal tubular function | Secondary hyperparathyroidism (of renal origin) Other specified disorders resulting from impaired renal function |
| N259 | 5889 | Disorder resulting from impaired renal tubular function, unspecified | Unspecified disorder resulting from impaired renal function |
| End Sta | To Done | I Disease (ESRD) Dx | |
| End-Stag<br>ICD10 | | ICD10 Description | ICD9 Description |
| I953 | | Hypotension of hemodialysis | Hypotension of hemodialysis |
| N185 | | Chronic kidney disease, stage 5 | Chronic kidney disease, Stage V |
| 11107 | ددەد | Cinomic Ridney disease, stage 3 | emone rancy disease, stage v |

| | 5056 | le i | |
|---|---|---|---|
| N186 | 5856 | End stage renal disease | End stage renal disease |
| T82818 | 99673 | Embolism due to vascular prosthetic devices, implants and | Other complications due to renal dialysis device, implant, and graft |
| A | 00650 | grafts, initial encounter | |
| T82828 | 99673 | Fibrosis due to vascular prosthetic devices, implants and grafts, initial encounter | Other complications due to renal dialysis device, implant, and graft |
| A<br>T82838 | 99673 | Hemorrhage due to vascular prosthetic devices, implants and | Other complications due to renal dialysis device, implant, and graft |
| 182838 | 990/3 | grafts, initial encounter | Other complications due to renai dialysis device, impiant, and graft |
| T82848 | 99673 | Pain due to vascular prosthetic devices, implants and grafts, | Other complications due to renal dialysis device, implant, and graft |
| A | 990/3 | initial encounter | Other complications due to renar dialysis device, implant, and grant |
| T82858 | 99673 | Stenosis of other vascular prosthetic devices, implants and | Other complications due to renal dialysis device, implant, and graft |
| A | 33073 | grafts, initial encounter | Other complications due to renar diarysis device, implant, and graft |
| T82868 | 99673 | Thrombosis due to vascular prosthetic devices, implants and | Other complications due to renal dialysis device, implant, and graft |
| A | 77013 | grafts, initial encounter | Other complications due to renar diarysis device, implant, and grant |
| T82898 | 99673 | Other specified complication of vascular prosthetic devices, | Other complications due to renal dialysis device, implant, and graft |
| A | ,,,,,, | implants and grafts, initial encounter | o their complications due to rotal diarysis device, implant, and grait |
| T85611 | 99656 | Breakdown (mechanical) of intraperitoneal dialysis catheter, | Mechanical complication due to peritoneal dialysis catheter |
| A | ,,,,,, | initial encounter | |
| T85621 | 99656 | Displacement of intraperitoneal dialysis catheter, initial | Mechanical complication due to peritoneal dialysis catheter |
| A | | encounter | |
| T85631 | 99656 | Leakage of intraperitoneal dialysis catheter, initial encounter | Mechanical complication due to peritoneal dialysis catheter |
| A | | | |
| T85691 | 99656 | Other mechanical complication of intraperitoneal dialysis | Mechanical complication due to peritoneal dialysis catheter |
| A | <u></u> | catheter, initial encounter | |
| T8571X | 99668 | Infection and inflammatory reaction due to peritoneal dialysis | Infection and inflammatory reaction due to peritoneal dialysis catheter |
| A | | catheter, initial encounter | |
| T8610 | | Unspecified complication of kidney transplant | Complications of transplanted kidney |
| T8611 | | Kidney transplant rejection | Complications of transplanted kidney |
| T8612 | | Kidney transplant failure | Complications of transplanted kidney |
| T8613 | | Kidney transplant infection | Complications of transplanted kidney |
| T8619 | | Other complication of kidney transplant | Complications of transplanted kidney |
| Z4822 | V420 | Encounter for aftercare following kidney transplant | Kidney replaced by transplant |
| Z4901 | V561 | Encounter for fitting and adjustment of extracorporeal dialysis | Fitting and adjustment of extracorporeal dialysis catheter |
| 7.1000 | X 7.5.60 | catheter | |
| Z4902 | V562 | Encounter for fitting and adjustment of peritoneal dialysis catheter | Fitting and adjustment of peritoneal dialysis catheter |
| Z4931 | V/5621 | Encounter for adequacy testing for hemodialysis | Encounter for adequacy testing for hemodialysis |
| Z4931 | V 3031 | Encounter for adequacy testing for hemodiarysis | Encounter for adequacy testing for hemodiarysis |
| Z4932 | V568 | Encounter for adequacy testing for peritoneal dialysis | Encounter for other dialysis |
| Z9115 | | Patient's noncompliance with renal dialysis | Noncompliance with renal dialysis |
| 2,110 | | a united the monetary manages with a united the same same same same same same same sam | Tronsompulation with rolling daily old |
| Z940 | V420 | Kidney transplant status | Kidney replaced by transplant |
| Z992 | | Dependence on renal dialysis | Renal dialysis status |
| | | ·r· ·· ·· ·· · | |
| End-Stag | ge Rena | l Disease (ESRD) Px | |
| | ICD9 | ICD10 Description | ICD9 Description |
| 03130JD | 3993 | Bypass Right Subclavian Artery to Upper Arm Vein with | Insertion of vessel-to-vessel cannula |
| | L | Synthetic Substitute, Open Approach | _ |
| 03130Z | 3927 | Bypass Right Subclavian Artery to Upper Arm Vein, Open | Arteriovenostomy for renal dialysis |
| D | | Approach | Arteriovenostomy for renal dialysis |
| | | Approach Bypass Left Subclavian Artery to Upper Arm Vein with | Arteriovenostomy for renal dialysis Insertion of vessel-to-vessel cannula |
| D<br>03140JD | 3993 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach | Insertion of vessel-to-vessel cannula |
| D<br>03140JD<br>03140Z | | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open | • • |
| D<br>03140JD<br>03140Z<br>D | 3993<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509 | 3993 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with | Insertion of vessel-to-vessel cannula |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V | 3993<br>3927<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A | 3993<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A<br>V | 3993<br>3927<br>3927<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A | 3993<br>3927<br>3927<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach Bypass Right Axillary Artery to Upper Arm Vein with | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A<br>V<br>03150JD | 3993<br>3927<br>3927<br>3927<br>3993 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach Bypass Right Axillary Artery to Upper Arm Vein with Synthetic Substitute, Open Approach | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Insertion of vessel-to-vessel cannula |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A<br>V | 3993<br>3927<br>3927<br>3927<br>3993 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach Bypass Right Axillary Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A<br>V<br>03150JD | 3993<br>3927<br>3927<br>3927<br>3993<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach Bypass Right Axillary Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A<br>V<br>03150JD<br>03150JV | 3993<br>3927<br>3927<br>3927<br>3993 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach Bypass Right Axillary Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Insertion of vessel-to-vessel cannula |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A<br>V<br>03150JD<br>03150JV | 3993<br>3927<br>3927<br>3927<br>3993<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach Bypass Right Axillary Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Nonautologous Tissue Substitute, Open Approach | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A<br>V<br>03150JD<br>03150JV<br>03150JV | 3993<br>3927<br>3927<br>3927<br>3993<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach Bypass Right Axillary Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Nonautologous Tissue Substitute, Open Approach Bypass Right Axillary Artery to Upper Arm Vein, Open | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A<br>V<br>03150JD<br>03150JV<br>03150JV<br>03150JV | 3993<br>3927<br>3927<br>3927<br>3993<br>3927<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach Bypass Right Axillary Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Nonautologous Tissue Substitute, Open Approach Bypass Right Axillary Artery to Upper Arm Vein, Open Approach | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis |
| D<br>03140JD<br>03140Z<br>D<br>031509<br>V<br>03150A<br>V<br>03150JD<br>03150JV<br>03150JV | 3993<br>3927<br>3927<br>3927<br>3993<br>3927 | Approach Bypass Left Subclavian Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Left Subclavian Artery to Upper Arm Vein, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Venous Tissue, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Autologous Arterial Tissue, Open Approach Bypass Right Axillary Artery to Upper Arm Vein with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Synthetic Substitute, Open Approach Bypass Right Axillary Artery to Superior Vena Cava with Nonautologous Tissue Substitute, Open Approach Bypass Right Axillary Artery to Upper Arm Vein, Open | Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis Insertion of vessel-to-vessel cannula Arteriovenostomy for renal dialysis Arteriovenostomy for renal dialysis |

| 031609 | 3927 | Bypass Left Axillary Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
|---|---|---|---|
| V | | Autologous Venous Tissue, Open Approach | |
| 03160A | 3927 | Bypass Left Axillary Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
| V | 3721 | Autologous Arterial Tissue, Open Approach | Tricolovenoscomy for renar diarysis |
| 021(010 | 2002 | | Y ( C 1 ( 1 1 1 |
| 03160JD | 3993 | Bypass Left Axillary Artery to Upper Arm Vein with | Insertion of vessel-to-vessel cannula |
| | | Synthetic Substitute, Open Approach | |
| 03160JV | 3927 | Bypass Left Axillary Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
| | | Synthetic Substitute, Open Approach | |
| 03160K | 3927 | Bypass Left Axillary Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
| | 3921 | | Arteriovenostomy for renai dialysis |
| V | | Nonautologous Tissue Substitute, Open Approach | |
| 03160Z | 3927 | Bypass Left Axillary Artery to Upper Arm Vein, Open | Arteriovenostomy for renal dialysis |
| D | | Approach | |
| 03160Z | 3927 | Bypass Left Axillary Artery to Superior Vena Cava, Open | Arteriovenostomy for renal dialysis |
| 03100Z | 3921 | | Afteriovenostomy for renar dialysis |
| V | | Approach | |
| 031709 | 3927 | Bypass Right Brachial Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
| V | | Autologous Venous Tissue, Open Approach | |
| 03170A | 3927 | Bypass Right Brachial Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
| V | 3721 | Autologous Arterial Tissue, Open Approach | Tricolovenoscomy for remar dualysis |
| 03170JD | 3993 | Bypass Right Brachial Artery to Upper Arm Vein with | Insertion of vessel-to-vessel cannula |
| | | Synthetic Substitute, Open Approach | |
| 03170JV | 3927 | Bypass Right Brachial Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
| | | Synthetic Substitute, Open Approach | |
| 03170K | 2027 | Bypass Right Brachial Artery to Superior Vena Cava with | A storiovanactamy for ranal dialysis |
| 031/0K | 3927 | | Arteriovenostomy for renal dialysis |
| V | <u></u> | Nonautologous Tissue Substitute, Open Approach | |
| 03170Z | 3927 | Bypass Right Brachial Artery to Upper Arm Vein, Open | Arteriovenostomy for renal dialysis |
| D | | Approach | |
| | 2027 | Bypass Right Brachial Artery to Superior Vena Cava, Open | Autoria annotana Communi Hallada |
| | 3927 | 1 ** * | Arteriovenostomy for renal dialysis |
| V | | Approach | |
| 031809 | 3927 | Bypass Left Brachial Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
| V | | Autologous Venous Tissue, Open Approach | |
| 03180A | 3927 | Bypass Left Brachial Artery to Superior Vena Cava with | A stariavanagtamy for sanal dialygic |
| 03180A | 3921 | | Arteriovenostomy for renal dialysis |
| V | | Autologous Arterial Tissue, Open Approach | |
| 03180JD | 3993 | Bypass Left Brachial Artery to Upper Arm Vein with | Insertion of vessel-to-vessel cannula |
| | | Synthetic Substitute, Open Approach | |
| 03180JV | 3027 | Bypass Left Brachial Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
| 031803 V | 3721 | | Arteriovenostomy for renar diarysis |
| | | Synthetic Substitute, Open Approach | |
| 03180K | 3927 | Bypass Left Brachial Artery to Superior Vena Cava with | Arteriovenostomy for renal dialysis |
| V | | Nonautologous Tissue Substitute, Open Approach | |
| 03180Z | 3927 | Bypass Left Brachial Artery to Upper Arm Vein, Open | Arteriovenostomy for renal dialysis |
| D | 3,2, | Approach | There is the state of the state |
| | | 11 | |
| 03180Z | 3927 | Bypass Left Brachial Artery to Superior Vena Cava, Open | Arteriovenostomy for renal dialysis |
| V | | Approach | |
| 03190JF | 3993 | Bypass Right Ulnar Artery to Lower Arm Vein with Synthetic | Insertion of vessel-to-vessel cannula |
| | | Substitute, Open Approach | |
| 0210075 | 2027 | | Autoria accordante Comunical distriction |
| 03190ZF | 3927 | Bypass Right Ulnar Artery to Lower Arm Vein, Open | Arteriovenostomy for renal dialysis |
| | | Approach | |
| 031A0J | 3993 | Bypass Left Ulnar Artery to Lower Arm Vein with Synthetic | Insertion of vessel-to-vessel cannula |
| F | | Substitute, Open Approach | |
| 031A0Z | 3027 | Bypass Left Ulnar Artery to Lower Arm Vein, Open | Arteriovenostomy for renal dialysis |
| USTAUZ | 394/ | 1 ** | Arteriovenostomy for renal dialysis |
| F | | Approach | |
| 031B0JF | 3994 | Bypass Right Radial Artery to Lower Arm Vein with | Replacement of vessel-to-vessel cannula |
| | | Synthetic Substitute, Open Approach | |
| 031B0Z | 3927 | Bypass Right Radial Artery to Lower Arm Vein, Open | Arteriovenostomy for renal dialysis |
| E OSTBOZ | 3741 | | Tricitovenosionily for reliar diarysis |
| L, | | Approach | |
| 031C0JF | 3994 | Bypass Left Radial Artery to Lower Arm Vein with Synthetic | Replacement of vessel-to-vessel cannula |
| | | Substitute, Open Approach | |
| 031C0Z | 3927 | Bypass Left Radial Artery to Lower Arm Vein, Open | Arteriovenostomy for renal dialysis |
| F | 3721 | Approach | 1.1.0.1.0.1.0.1.0.1.1.1.1.1.1.1.1.1.1.1 |
| | 20.75 | | In the second second |
| 03LK0C | 3953 | Occlusion of Right Internal Carotid Artery with Extraluminal | Repair of arteriovenous fistula |
| Z | | Device, Open Approach | |
| 03LK0Z | 3953 | Occlusion of Right Internal Carotid Artery, Open Approach | Repair of arteriovenous fistula |
| 7 | 1220 | The state of the s | · <u>*</u> · |
| 021 772 6 | 2052 | O I CONTINUE TO STATE OF THE CONTINUE TO STATE | |
| 03LK3C | 3953 | Occlusion of Right Internal Carotid Artery with Extraluminal | Repair of arteriovenous fistula |
| Z | <u> </u> | Device, Percutaneous Approach | |
| 03LK3Z | 3953 | Occlusion of Right Internal Carotid Artery, Percutaneous | Repair of arteriovenous fistula |
| Z | | Approach | _ ^ |
| . — | 1 | rr ····· | 1 |

| · . | | | |
|---|---|---|---|
| 03LK4C<br>Z | 3953 | Occlusion of Right Internal Carotid Artery with Extraluminal Device, Percutaneous Endoscopic Approach | Repair of arteriovenous fistula |
| 03LK4Z<br>Z | 3953 | Occlusion of Right Internal Carotid Artery, Percutaneous Endoscopic Approach | Repair of arteriovenous fistula |
| 03LL0C | 3953 | Occlusion of Left Internal Carotid Artery with Extraluminal | Repair of arteriovenous fistula |
| 03LL0Z<br>Z | 3953 | Device, Open Approach Occlusion of Left Internal Carotid Artery, Open Approach | Repair of arteriovenous fistula |
| 03LL3C<br>Z | 3953 | Occlusion of Left Internal Carotid Artery with Extraluminal Device, Percutaneous Approach | Repair of arteriovenous fistula |
| 03LL3Z<br>Z | 3953 | Occlusion of Left Internal Carotid Artery, Percutaneous<br>Approach | Repair of arteriovenous fistula |
| 03LL4C<br>Z | 3953 | Occlusion of Left Internal Carotid Artery with Extraluminal Device, Percutaneous Endoscopic Approach | Repair of arteriovenous fistula |
| 03LL4Z<br>Z | 3953 | Occlusion of Left Internal Carotid Artery, Percutaneous Endoscopic Approach | Repair of arteriovenous fistula |
| 03PY07<br>Z | 3943 | * ** | Removal of arteriovenous shunt for renal dialysis |
| 03PY0J<br>Z | 3994 | Removal of Synthetic Substitute from Upper Artery, Open<br>Approach | Replacement of vessel-to-vessel cannula |
| 03PY0K<br>Z | 3943 | Removal of Nonautologous Tissue Substitute from Upper<br>Artery, Open Approach | Removal of arteriovenous shunt for renal dialysis |
| 03PY37<br>Z | 3943 | | Removal of arteriovenous shunt for renal dialysis |
| 03PY3J<br>Z | 3994 | Removal of Synthetic Substitute from Upper Artery,<br>Percutaneous Approach | Replacement of vessel-to-vessel cannula |
| 03PY3K<br>Z | 3943 | Removal of Nonautologous Tissue Substitute from Upper<br>Artery, Percutaneous Approach | Removal of arteriovenous shunt for renal dialysis |
| 03PY47<br>Z | 3943 | Removal of Autologous Tissue Substitute from Upper Artery,<br>Percutaneous Endoscopic Approach | Removal of arteriovenous shunt for renal dialysis |
| 03PY4J<br>Z | 3994 | Removal of Synthetic Substitute from Upper Artery,<br>Percutaneous Endoscopic Approach | Replacement of vessel-to-vessel cannula |
| 03PY4K<br>Z | 3943 | Removal of Nonautologous Tissue Substitute from Upper<br>Artery, Percutaneous Endoscopic Approach | Removal of arteriovenous shunt for renal dialysis |
| 03VK0C<br>Z | 3953 | | Repair of arteriovenous fistula |
| 03VK3C<br>Z | 3953 | | Repair of arteriovenous fistula |
| 03VK4C<br>Z | 3953 | Restriction of Right Internal Carotid Artery with Extraluminal Device, Percutaneous Endoscopic Approach | Repair of arteriovenous fistula |
| 03VL0C<br>Z | 3953 | Restriction of Left Internal Carotid Artery with Extraluminal<br>Device, Open Approach | Repair of arteriovenous fistula |
| 03VL3C<br>Z | 3953 | Restriction of Left Internal Carotid Artery with Extraluminal Device, Percutaneous Approach | Repair of arteriovenous fistula |
| 03VL4C<br>Z | 3953 | Restriction of Left Internal Carotid Artery with Extraluminal<br>Device, Percutaneous Endoscopic Approach | Repair of arteriovenous fistula |
| 03WY0J<br>Z | 3994 | Revision of Synthetic Substitute in Upper Artery, Open<br>Approach | Replacement of vessel-to-vessel cannula |
| 03WY3J<br>Z | 3994 | Revision of Synthetic Substitute in Upper Artery,<br>Percutaneous Approach | Replacement of vessel-to-vessel cannula |
| 03WY4J<br>Z | | Revision of Synthetic Substitute in Upper Artery,<br>Percutaneous Endoscopic Approach | Replacement of vessel-to-vessel cannula |
| 03WYX<br>JZ | | Revision of Synthetic Substitute in Upper Artery, External<br>Approach | Replacement of vessel-to-vessel cannula |
| 05HY33<br>Z | | Insertion of Infusion Device into Upper Vein, Percutaneous Approach | Venous catheterization for renal dialysis |
| 06HY33<br>Z | | Insertion of Infusion Device into Lower Vein, Percutaneous Approach | Venous catheterization for renal dialysis |
| 0TS00Z<br>Z | | Reposition Right Kidney, Open Approach | Renal autotransplantation |
| Z | 5561 | Reposition Left Kidney, Open Approach | Renal autotransplantation |
| 0TY00Z<br>0 | | | Other kidney transplantation |
| 0TY00Z<br>1 | 5569 | Transplantation of Right Kidney, Syngeneic, Open Approach | Other kidney transplantation |

| 0TY00Z<br>2 | 5569 | Transplantation of Right Kidney, Zooplastic, Open Approach | Other kidney transplantation |
|---|---|---|---|
| 0TY10Z<br>0 | 5569 | Transplantation of Left Kidney, Allogeneic, Open Approach | Other kidney transplantation |
| 0TY10Z<br>1 | 5569 | Transplantation of Left Kidney, Syngeneic, Open Approach | Other kidney transplantation |
| 0TY10Z<br>2 | 5569 | Transplantation of Left Kidney, Zooplastic, Open Approach | Other kidney transplantation |
| 3E1M39<br>Z | 5498 | Irrigation of Peritoneal Cavity using Dialysate, Percutaneous<br>Approach | Peritoneal dialysis |
| 5A1D70<br>Z | | Performance of Urinary Filtration, Intermittent, Less than 6<br>Hours Per Day | Hemodialysis |
| 5A1D80<br>Z | | Performance of Urinary Filtration, Prolonged Intermittent, 6-<br>18 hours Per Day | Hemodialysis |
| 5A1D90<br>Z | 3995 | Performance of Urinary Filtration, Continuous, Greater than<br>18 hours Per Day | Hemodialysis |
| Heart Fai | ilure Dx | | |
| ICD10 | ICD9 | ICD10 Description | ICD9 Description |
| 10981 | | Rheumatic heart failure | Rheumatic heart failure (congestive) |
| I110 | | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| I110<br>I130 | | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and with |
| | | failure and stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | chronic kidney disease stage I through stage IV, or unspecified |
| I132 | 40493 | Hypertensive heart and chronic kidney disease with heart failure and with stage 5 chronic kidney disease, or end stage renal disease | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and chronic kidney disease stage V or end stage renal disease |
| I501 | 4281 | Left ventricular failure, unspecified | Left heart failure |
| 15020 | | Unspecified systolic (congestive) heart failure | Congestive heart failure, unspecified |
| 15021 | 4280 | Acute systolic (congestive) heart failure | Congestive heart failure, unspecified |
| 15022 | | Chronic systolic (congestive) heart failure | Congestive heart failure, unspecified |
| I5023 | 4280 | Acute on chronic systolic (congestive) heart failure | Congestive heart failure, unspecified |
| I5030 | | Unspecified diastolic (congestive) heart failure | Congestive heart failure, unspecified |
| I5031 | | Acute diastolic (congestive) heart failure | Congestive heart failure, unspecified |
| I5032 | 4280 | Chronic diastolic (congestive) heart failure | Congestive heart failure, unspecified |
| I5033 | 4280 | Acute on chronic diastolic (congestive) heart failure | Congestive heart failure, unspecified |
| I5040 | 4280 | Unspecified combined systolic (congestive) and diastolic (congestive) heart failure | Congestive heart failure, unspecified |
| I5041 | | Acute combined systolic (congestive) and diastolic (congestive) heart failure | Congestive heart failure, unspecified |
| I5042 | | Chronic combined systolic (congestive) and diastolic (congestive) heart failure | Congestive heart failure, unspecified |
| I5043 | | (congestive) heart failure | Congestive heart failure, unspecified |
| I50810 | | Right heart failure, unspecified | Heart failure, unspecified |
| I50811 | | Acute right heart failure | Heart failure, unspecified |
| I50812 | 4289 | Chronic right heart failure | Heart failure, unspecified |
| I50813 | 4289 | Acute on chronic right heart failure | Heart failure, unspecified |
| I50814 | 4280 | Right heart failure due to left heart failure | Congestive heart failure, unspecified |
| I5082 | 4289 | Biventricular heart failure | Heart failure, unspecified |
| I5083 | 4289 | High output heart failure | Heart failure, unspecified |
| I5084 | | End stage heart failure | Heart failure, unspecified |
| 15089 | 4289 | Other heart failure | Heart failure, unspecified |
| 1509 | | Heart failure, unspecified | Heart failure, unspecified |
| | | rroute randre, unspecified | rrout randre, anapoented |
| Hypotens | | ICD10 Days 2 of the | TCD0 D |
| | | ICD10 Description | ICD9 Description |
| 1950 | | Idiopathic hypotension | Chronic hypotension |
| I951 | | Orthostatic hypotension | Orthostatic hypotension |
| I953 | | Hypotension of hemodialysis | Hypotension of hemodialysis |
| I9589 | | Other hypotension | Other specified hypotension |
| 1959 | | Hypotension, unspecified | Hypotension, unspecified |
| 1952 | 45829 | Hypotension due to drugs | Other iatrogenic hypotension |
| 19581 | | Postprocedural hypotension | Other iatrogenic hypotension |
| Hyperkal | | , ,, | · |
| | | ICD10 Description | ICD9 Description |
| E875 | | Hyperkalemia | Hyperpotassemia |
| 2010 | 2,01 | J P v · | ***JP**Pomooviiiu |